CLINICAL TRIAL: NCT02777099
Title: Impact of Remote Ischemic Postconditioning on Autonomic Function and Prognosis in Clients With Acute Ischemic Stroke
Brief Title: Impact of Remote Ischemic Postconditioning on Autonomic Function in Stroke Patients
Acronym: IRAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014A020212455
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Ischemic Stroke
Keywords: remote ischemic postconditioning; autonomic function; heart rate variability; acute ischemic stroke; prognosis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RIPostC (Experimental): Receiving RIPostC with pressure set at 200 mmHg. Intervention:Procedure:Remote Ischemic Postconditioning
  Interventions: Procedure: remote ischemic postconditioning
- sham RIPostC (Sham Comparator): Receiving sham RIPostC with pressure set at the patient's diastolic blood pressure.
  Intervention:Procedure:Sham Remote Ischemic Postconditioning
  Interventions: Procedure: sham remote ischemic postconditioning

INTERVENTIONS:
Procedure: remote ischemic postconditioning — Remote ischemic postconditioning was performed by 4 cycles of upper-limb ischemia and reperfusion.The upper-limb ischemia was induced by inflating a blood pressure cuff on a healthy upper arm to 200 mmHg for 5 min,and then deflating it for 5 min.Each patients in the PIPostC group will have the treatment once a day for 30 days.
  Other Names: PIPostC
  Arms: RIPostC
Procedure: sham remote ischemic postconditioning — Sham remote ischemic postconditioning was performed by 4 cycles of upper-limb ischemia and reperfusion. The upper-limb ischemia was induced by inflating a blood pressure cuff on a healthy upper arm to the patient's actual diastolic blood pressure for 5 min,and then deflating it for 5 min.Each patients in the sham PIPostC group will have the sham treatment once a day for 30 days.
  Other Names: sham PIPostC
  Arms: sham RIPostC

SUMMARY:
The purpose of this study is to determine whether remote ischemic postconditioning (RIPostC) initiates autonomic nervous system response and affects the prognosis in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
Remote ischemic postconditioning (RIPostC) has proven effective in reducing the ischemia-reperfusion injury. But the defensive mechanism of RIPostC still unclear. Stroke is frequently associated with autonomic dysfunction. Heart rate variability (HRV) represents the autonomic nervous system activity.This study aims to investigate whether RIPostC correlates with autonomic function and thus predicts prognosis of stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as ischemic stroke according to the Chinese guideline of diagnosis and treatment of acute ischemic stroke 2010
2. Age between 18 to 85 years old
3. initial ischemic stroke within 14 days or less.
4. National Institutes of Health Stroke Scale (NIHSS)score 0-15
5. Modified Rankin Scale(mRS)score 1-4
6. Informed consent

Exclusion Criteria:

1. Intravenous or arterial thrombolysis, or revascularization
2. Acute myocardial infarction,atrial fibrillation,arrhythmia,or cardiogenic cerebral embolism
3. Systolic Blood Pressure(SBP)>200mmHg after medication treatment
4. Plasma fibrinogen>7g/L
5. Upper limb fracture or percutaneous injury
6. Subclavian artery stenosis
7. With severe cardiac,respiratory,hepatic,and renal dysfunction or malignant tumor
8. Simultaneous participation in another interventional study
9. Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-02 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variabilities | at the time points of baseline and 7 and 30 days after treatments
  Heart rate variability (HRV) is one of the most promising markers represent for autonomic function.We assess the changes from baseline heart rate variability to 7days and 30days.

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale(NIHSS) | at the time points of baseline and 7days after treatments.
  National Institutes of Health Stroke Scale(NIHSS)is a commonly used scale for quantifing the impairment caused by a stroke objectively.
Modified Rankin scale(mRS) | at the time points of baseline and 7,30 and 90 days after treatments
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.The scale runs from 0-6, running from perfect health without symptoms to death.0 - No symptoms.1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3 - Moderate disability. Requires some help, but able to walk unassisted.4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.6 - Dead.
Barthel Index(BI) | at the time points of baseline and 7,30 and 90 days after treatments
  The Barthel Index scale is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking.It uses ten variables describing ADL and mobility. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital.The ten variables addressed in the Barthel scale are:presence or absence of fecal incontinence;presence or absence of urinary incontinence;help needed with grooming;help needed with toilet use help needed with feeding;help needed with transfers (e.g. from chair to bed) help needed with walking;help needed with dressing;help needed with climbing stairs;and help needed with bathing.

OTHER OUTCOMES:
Stroke Recurrence | 90 days after treatments
  Stroke recurrence is commonly used to estimate the prognosis of stroke.
Mortality | 90 days after treatments
  Mortality is commonly used to estimate the prognosis of stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Lin WEI, MD, Study Chair — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liang H, Ye R, Zhang X, Ye H, Ouyang W, Cai S, Wei L. Autonomic function may mediate the neuroprotection of remote ischemic postconditioning in stroke: A randomized controlled trial. J Stroke Cerebrovasc Dis. 2023 Aug;32(8):107198. doi: 10.1016/j.jstrokecerebrovasdis.2023.107198. Epub 2023 Jun 15. PMID 37329785